CLINICAL TRIAL: NCT01223261
Title: Observational Study of Surgical Treatment of Necrotizing Enterocolotis or Isolated Intestinal Perforation
Brief Title: Observational Study of Surgical Treatment of Necrotizing Enterocolotis
Acronym: NEC Surgery
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Martin L. Blakely, Lead Principal Investigator, University of Texas Health Science Center at Houston
Other Study IDs: NICHD-NRN-0027; U10HD034216 (NIH); U10HD027904 (NIH); U10HD021364 (NIH); M01RR000080 (NIH); U10HD027853 (NIH); M01RR008084 (NIH); U10HD027851 (NIH); M01RR000039 (NIH); U10HD021397 (NIH); M01RR016587 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); U10HD027880 (NIH); M01RR000070 (NIH); U10HD040689 (NIH); M01RR000633 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); M01RR006022 (NIH); U10HD040492 (NIH); M01RR000030 (NIH); U10HD040498 (NIH); M01RR007122 (NIH); U10HD040521 (NIH); M01RR000044 (NIH); U10HD040461 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Enterocolitis, Necrotizing; Intestinal Perforation
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Laparotomy; Drainage; Isolated intestinal perforation; Focal intestinal performation
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing; Intestinal Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purposes of this study were: 1) to compare mortality and postoperative morbidities in extremely low birth weight (ELBW) infants who underwent initial laparotomy or drainage for necrotizing enterocolitis (NEC) or isolated intestinal perforation (IP); 2) to determine the ability to distinguish NEC from IP preoperatively and the importance of this distinction on outcome measures; and 3) to evaluate the association between extent of intestinal disease determined at operation and outcome measures. All ELBW infants born at participating NRN centers were screened for the presence of NEC or IP that was thought by the pediatric surgeon and neonatologist to require surgical intervention. Data were collected enrolled infants, including: intraoperative findings recorded by the surgeon and specific post-operative complications. Neurodevelopmental examinations were conducted on surviving infants at 18-22 months corrected age.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is a condition, generally affecting premature infants, in which the intestines become ischemic (lack oxygen and/or blood flow). NEC occurs in up to 5-15% of extremely low birth weight (ELBW) infants. Isolated or focal intestinal perforation (IP) is a less common condition, affecting an estimated 4% of ELBWs, in which a hole develops in the intestines leaking fluid into the abdomin. The outcomes for infants with NEC or IP are poor: 49% die and half of the surviving infants are neurodevelopmentally impaired.

Surgical options for NEC and IP include two possible procedures: peritoneal drainage, in which a tube is placed in the abdominal cavity through a small incision for fluid to drain out; or laparotomy, in which an incision is made in the abdomen and diseased intestine is removed. Infants treated with an initial drainage sometimes go on to need a laparotomy. Most surgeons now believe that a diagnosis of the intestinal perforation (IP) may actually be either true NEC or a different and distinct pathology, termed isolated intestinal perforation. The ability to distinguish these 2 conditions preoperatively, based on perinatal characteristics, physical examination findings, and findings on abdominal plain film imaging, remains unknown. If these 2 entities can be distinguished preoperatively, the intervention chosen and outcomes may be different. From the two available surgical options, tt is not known whether initial laparotomy or peritoneal drain placement is more effective for either NEC or IP.

This study was a prospective, multicenter observational study to describe the surgical outcomes (mortality, post-operative intestinal stricture, intra-abdominal abscess formation, etc.) in ELBW infants with either NEC or IP who underwent initial laparotomy or peritoneal drainage. We also evaluated the ability of surgeons to distinguish NEC and IP pre-operatively and the relevance of this distinction on outcome. Finally, an analysis of the impact of extent of intestinal involvement with NEC on outcome measures is reported.

All ELBW infants born at participating NRN centers were screened for the presence of NEC or IP that was thought by the pediatric surgeon and neonatologist to require surgical intervention. Data were collected enrolled infants, including: intraoperative findings recorded by the surgeon and specific post-operative complications.

Neurodevelopmental examinations were conducted on surviving infants at 18-22 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born 401-1,000 grams at birth enrolled in the NRN Generic Database
* Sage III NEC or isolated intestinal perforation
* Pediatric surgeon decision to perform surgery for suspected NEC or IP

Exclusion Criteria:

* Decision not to treat

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely Low Birth Weight (ELBW) infants (those with birth weights <1000 g) born at participating NRN Centers diagnosed by a pediatric surgeon and neonatologist as having either necrotizing enterocolitis (NEC) or intestinal perforation (IP) requiring surgical intervention.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2001-03; Primary Completion 2002-09 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a randomized trial | 1 year
  Ability to enroll infants in a 1-year period

SECONDARY OUTCOMES:
Document variation in current surgical practices | Until hospital discharge or 120 days of life
Prevalence of infants who would qualify for the study | Until hospital discharge or 120 days of life
Frequency of postoperative complications | Until hospital discharge or 120 days of life
Neurodevelopmental impairment | 18-22 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Martin L. Blakely, MD, Study Director — The University of Texas Health Science Center, Houston; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies & Children's Hospital; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; Charles R. Bauer, MD, Principal Investigator — University of Miami; James A. Lemons, MD, Principal Investigator — Indiana University; David K. Stevenson, MD, Principal Investigator — Stanford University; Abbot R. Laptook, MD, Principal Investigator — University of Texas; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Ronald N. Goldberg, MD, Principal Investigator — Duke University; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; W. Kenneth Poole, PhD, Principal Investigator — RTI International
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Result] Blakely ML, Lally KP, McDonald S, Brown RL, Barnhart DC, Ricketts RR, Thompson WR, Scherer LR, Klein MD, Letton RW, Chwals WJ, Touloukian RJ, Kurkchubasche AG, Skinner MA, Moss RL, Hilfiker ML; NEC Subcommittee of the NICHD Neonatal Research Network. Postoperative outcomes of extremely low birth-weight infants with necrotizing enterocolitis or isolated intestinal perforation: a prospective cohort study by the NICHD Neonatal Research Network. Ann Surg. 2005 Jun;241(6):984-9; discussion 989-94. doi: 10.1097/01.sla.0000164181.67862.7f. PMID 15912048
- [Result] Blakely ML, Tyson JE, Lally KP, McDonald S, Stoll BJ, Stevenson DK, Poole WK, Jobe AH, Wright LL, Higgins RD; NICHD Neonatal Research Network. Laparotomy versus peritoneal drainage for necrotizing enterocolitis or isolated intestinal perforation in extremely low birth weight infants: outcomes through 18 months adjusted age. Pediatrics. 2006 Apr;117(4):e680-7. doi: 10.1542/peds.2005-1273. Epub 2006 Mar 20. PMID 16549503
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/